CLINICAL TRIAL: NCT05461911
Title: Prospective Multicenter Randomized Controlled Low-interventional Post-registration Study to Assess the Clinical Efficacy of the Specialized Enteral Tube Nutrition Composition Nutrison Advanced Cubison as a Part of Complex Pressure Ulcers (PU) Therapy Versus Standard Enteral Tube Nutrition Products
Brief Title: Study to Assess the Clinical Efficacy of the Specialized Enteral Tube Nutrition Composition Nutrison Advanced Cubison as a Part of Complex Pressure Ulcers (PU) Therapy
Status: Completed | Type: Observational
Sponsor: Enrollme.ru, LLC (Network)
Collaborators: Danone Nutricia (Industry)
Responsible Party: Sponsor
Other Study IDs: DECUBISON
Record Dates: First submitted 2022-07-12; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Pressure Ulcer ( Stage 2-3)
Keywords: Stroke; Traumatic Brain Injury
MeSH Terms: conditions — Pressure Ulcer; Stroke; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Study Group: 30 adult patients aged 30-75 years to receive a specialized tube feeding product Nutrison Advanced Cubison (20% protein energy 100 kcal, 5.5 g protein, 0.85 g arginine, 38 mg of vitamin C and 2 mg of zinc) in a volume not exceeding 1.5 liters / day and, if necessary, to replenish nutritional needs based on the total daily intake of 30-35 kcal / kg / day and 1.2-1.5 g of protein / kg body weight / day according to the recommendations for nutritional support for patients with pressure ulcers during the entire observation period
  Interventions: Dietary Supplement: Nutrison Advanced Cubison
- The Control Group: 30 patients aged 30-75 years to receive a standard (available in the clinic) tube feeding product (energetically similar to the product in group 1) with a standard content of arginine, vitamins and minerals from calculating the total daily intake of 30-35 kcal / kg / day and 1.2-1.5 g protein / kg body weight / day according to the recommendations for nutritional support for patients with pressure ulcers during the entire observation period

INTERVENTIONS:
Dietary Supplement: Nutrison Advanced Cubison — (20% protein energy 100 kcal, 5.5 g protein, 0.85 g arginine, 38 mg of vitamin C and 2 mg of zinc) in a volume not exceeding 1.5 liters / day and, if necessary, to replenish nutritional needs based on the total daily intake of 30-35 kcal / kg / day and 1.2-1.5 g of protein / kg body weight / day according to the recommendations for nutritional support
  Groups: The Study Group

SUMMARY:
A large number of studies are devoted to studying the effect of patient nutrition on the occurrence and treatment of pressure ulcers. Several studies, including the US National Long-term Treatment of Pressure Ulcers Study, have shown that weight loss and malnutrition were associated with a higher risk of pressure ulcers.

One of the successful products specially created for the treatment of pressure ulcers and taking into account the results of research is the high-protein, energy-rich, ready-to-use enteral tube feeding food product Nutrison Advanced Cubison. It is a complete enteral nutritional supplement with an innovative nutrient composition for patients with chronic wounds, including pressure ulcers, or at increased risk of developing them.

Taking into account the available data, it seems expedient to continue studying the unique combination of nutrients that make up the study food product Nutrison Advanced Cubison in order to develop the most effective nutritional protocols for patients at risk for the treatment and prevention of pressure ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with stroke / TBI and who are on tube feeding
* Presence of pressure ulcers of 2-3 stages
* Informed voluntary consent to medical intervention is formalized in accordance with the requirements of the Federal Law of 21.11.2011 N 323-FZ "On the basics of protecting the health of citizens in the Russian Federation."

Exclusion Criteria:

* Hemodynamically unstable patients
* Severe renal impairment (GFR <30 ml / min)
* Moderate or severe liver failure (Child-Pugh Class B or C)
* Oncological diseases (lasting more than 5 years)
* Hypersensitivity to any component of the test food mixture
* Inclusion in clinical interventional research
* Uncertainty of the investigator about the willingness or ability of the subject to comply with the protocol requirements
* Any other medical or non-medical reasons that, in the opinion of the physician, may prevent the patient from participating in the study

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients hospitalized with strokes or traumatic brain injury, who are on tube feeding and with the presence of pressure ulcers of 2-3 stages identified at baseline or during hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in the area of pressure ulcers in both groups during the study | up to 4 weeks
The proportion of patients in both groups with a decrease in the area of the pressure ulcer by 20% or more by the date of completion of observations | up to 4 weeks
Changes in the Pressure Ulcer Scale for Healing values in both groups during the study | up to 4 weeks
  Pressure Ulcer Scale for Healing (PUSH) is a common tool to monitor pressure healing over time. The PUSH Tool monitors three parameters: surface area of the wound, wound exudate and type of wound tissue. Minimum value is 0, maximum value is 17. The bigger scale is the worse

SECONDARY OUTCOMES:
Duration of treatment for pressure ulcers in study patients | up to 4 weeks
Frequency and duration of infectious complications of pressure ulcers in study patients | up to 4 weeks
Concentration of the blood albumin at the beginning and at the end of observations | up to 4 weeks
Concentration of the blood lymphocytes at the beginning and at the end of observations | up to 4 weeks
Concentration of the C-reactive protein at the beginning and at the end of observations | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Getman, Dr, Study Director — Enrollme.ru, LLC
Locations (3):
- Russia (3):
  - GAUZ Bryansk city hospital №1, Bryansk
  - GBUZ GKB named after VV Vinogradov DZM, Moscow
  - Hospital named after V.D. Seredavin, Samara

IPD SHARING:
Plan to Share IPD: Undecided